CLINICAL TRIAL: NCT04524598
Title: Limbix Spark: A CBT-based Mobile Intervention as First Line Treatment for Adolescent Depression During COVID-19
Brief Title: A CBT-based Mobile Intervention as First Line Treatment for Adolescent Depression During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Limbix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Limbix Spark 02
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Depression
Keywords: Adolescence; Digital Therapeutic; Cognitive Behavioral Therapy; Behavioral Activation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Limbix Spark (Experimental): A 5 week CBT-based intervention
  Interventions: Device: Limbix Spark
- Psychoeducation (Active Comparator): 5 weeks of psychoeducation about depression. Upon completion, participants will be automatically enrolled into the Limbix Spark CBT-based intervention
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Device: Limbix Spark — The Limbix Spark program is divided into 5 levels. Each level provides educational information about cognitive behavioral therapy and interactive activities.
  Arms: Limbix Spark
Other: Psychoeducation — The Psychoeducation program is divided into 5 lessons. Each lesson covers a different topic about depression.
  Arms: Psychoeducation

SUMMARY:
Over 3 million teenagers in the USA have depression, and rates of depression and suicide are sharply increasing. Teenage depression has far-reaching consequences including impairments in academic and work performance and social and family relationships, substance abuse, and worsening of other health conditions, which can persist into adulthood. Access to mental health care for teenagers is limited due to a shortage of mental health providers and many teenagers and parents are reluctant to take antidepressants. COVID-19 and mandated physical and social distancing is expected to increase rates of teenage depression, and further limit access to traditional methods of care (e.g. psychotherapy). This highlights an urgent need to develop accessible, digital treatments for teenage depression to address the serious mental health impacts of the COVID-19 pandemic. This fully virtual study (https://www.limbix.com/spark) will compare the relative safety, effectiveness, and engagement of a mobile application based on cognitive behavioral therapy and behavioral activation (Limbix Spark), focusing on the idea that engaging in behaviors that are rewarding or provide a sense of mastery can be effective in reducing symptoms of depression. Limbix Spark will be compared to a mobile app containing educational material about depression (Psychoeducation).

DETAILED DESCRIPTION:
Depression in adolescence is a public health crisis, with incidence and suicide rates rising sharply over the past decade. The COVID-19 global pandemic, along with mandated social and physical distancing, is expected to have substantial repercussions on public mental health and exacerbate the mental health crisis among teens. Adolescents, a group with significant unmet mental health needs, are at risk during this time, as they are especially vulnerable to depression and suicidality following environmental stressors, trauma, and social isolation that are endemic to this global pandemic. With difficulties in receiving in person care magnified during social distancing, now more than ever, there is an immediate need for safe, accessible, and effective digital treatments for mental health disorders.

The proposed intervention is intended to increase access to mental health care during the COVID-19 pandemic. This study aims to evaluate the clinical effectiveness and safety of a cognitive behavioral therapy (CBT)- based digital treatment for adolescent depression (Limbix Spark) relative to psychoeducation. Limbix Spark implements behavioral activation (BA), a key CBT skill that provides a sense of pleasure or mastery through self-monitored activities to reduce depressive symptoms and improve functional outcomes.

Adolescents with depression (13-21 years old) across the country will be recruited to participate in a fully remote, clinical trial via https://www.limbix.com/spark. At an initial virtual visit, following informed consent, adolescents and parents (for those under 18) will fill out standardized questionnaires designed to measure symptoms of depression, anxiety, and general health. Participants will then download an app onto their mobile phone and be randomly assigned to one of two groups. One group will receive the Limbix Spark program and the other will receive the Psychoeducation program for 5 weeks. The Limbix Spark program is divided into 5 levels. Each level provides educational information about cognitive behavioral therapy and behavioral activation, and interactive activities including mood tracking and activity scheduling. The Psychoeducation program is divided into 5 lessons. Each lesson covers a different topic about depression. During both 5 week programs, patients will also complete a weekly Patient Health Questionnaire, which is designed to measure depressive symptoms and also will report any negative side effects they may be experiencing. After 5 weeks, participants and legal guardians (for those under 18) will complete another set of standardized questionnaires designed to measure symptoms of depression, anxiety, and general health. Patients will also complete questionnaires asking them about their thoughts and experiences with the program they just completed. Lastly, a subset of patients and parents will be invited to complete a virtual interview to provide feedback on using the program.

The trial will be divided into two phases. The first phase will enroll 60 participants and participants will be randomized to either Spark and Control groups as described above. The second phase will enroll 175 participants and those randomized into the control group will be given access to the 5-week Spark intervention after completing the 5 weeks of control condition (control extension arm). Once completing the control extension arm, participants will complete a second set of post study questionnaires after 5 weeks.

All study participants that complete the 5-week Limbix Spark program and the post study questionnaires will be contacted and asked to consent to participation in the follow-up study. Only participants who did not opt-out to being contacted for future research will be contacted. This study will collect questionnaires from participants at any or all of the following time frames as indicated: 1-month, 3-month, and 6-month following completion of the Spark arm.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 13 and 21
* Self-reported symptoms of depression
* Will be residing in the USA for the duration of the 5-week study
* Under the care of a US-based primary care and/or licensed mental healthcare provider and willing and able to provide the name and contact information of the provider during consent appointment.
* English fluency and literacy of adolescent and consenting legal guardian if under 18
* Access to a smartphone (iPhone 5s or later or running Android 4.4 KitKat or later) and regular internet access
* Willing to provide informed e-consent/assent and have legal guardian willing to provide informed e-consent if under 18.

Exclusion Criteria:

* Self-reported lifetime suicide attempt or active self-harm or active suicidal ideation with intent
* Have a diagnosis by a clinician of bipolar disorder, substance use disorder, or any psychotic disorder including schizophrenia
* Incapable of understanding or completing study procedures and digital intervention as determined by participant, patient/legal guardian, healthcare provider, or clinical research team

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 227 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2022-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lake, PhD, Principal Investigator — Director of Research; Aarthi Padmanabhan, Phd, Principal Investigator — Research Director
Locations (1):
- Limbix Health, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peake E, Miller I, Flannery J, Chen L, Lake J, Padmanabhan A. Preliminary Efficacy of a Digital Intervention for Adolescent Depression: Randomized Controlled Trial. J Med Internet Res. 2024 Feb 7;26:e48467. doi: 10.2196/48467. PMID 38324367
- [Derived] Kulikov VN, Crosthwaite PC, Hall SA, Flannery JE, Strauss GS, Vierra EM, Koepsell XL, Lake JI, Padmanabhan A. A CBT-based mobile intervention as an adjunct treatment for adolescents with symptoms of depression: a virtual randomized controlled feasibility trial. Front Digit Health. 2023 May 23;5:1062471. doi: 10.3389/fdgth.2023.1062471. eCollection 2023. PMID 37323125

RESULTS

PARTICIPANT FLOW:
Groups:
- Limbix Spark - Phase I; Limbix Spark - Phase II: A 5 week CBT-based intervention
  Limbix Spark: The Limbix Spark program is divided into 5 levels. Each level provides educational information about cognitive behavioral therapy and interactive activities.
- Psychoeducation - Phase I; Psychoeducation - Phase II: 5 weeks of psychoeducation about depression. Upon completion, participants will be automatically enrolled into the Limbix Spark CBT-based intervention
  Psychoeducation: The Psychoeducation program is divided into 5 lessons. Each lesson covers a different topic about depression.
- Control Extension - Phase II: Participants who were initially assigned to the Psychoeducation control arm were given the opportunity to then complete the 5 week CBT-based intervention, Limbix Spark.
  Limbix Spark: The Limbix Spark program is divided into 5 levels. Each level provides educational information about cognitive behavioral therapy and interactive activities.
Period: Phase I - Feasibility
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation - Phase II | Control Extension - Phase II
Started | 35 | 25 | 0 | 0 | 0
Completed | 31 | 20 | 0 | 0 | 0
Not Completed | 4 | 5 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 4 | 0 | 0 | 0
Not completed — Dropped for missing two consecutive weekly safety check-ins. | 2 | 1 | 0 | 0 | 0
Period: Phase II - Outcomes
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation - Phase II | Control Extension - Phase II
Started | 0 | 0 | 80 | 80 | 0
Met PHQ-8 Threshold (Baseline >/= 10) (Participants who met this threshold were included in the intention-to-treat analysis and the per protocol analyses.) | 0 | 0 | 63 | 58 | 0
Completed | 0 | 0 | 54 | 67 | 0
Not Completed | 0 | 0 | 26 | 13 | 0
Not completed — Lost to Follow-up | 0 | 0 | 16 | 8 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0
Not completed — Dropped for missing two consecutive weekly safety check-ins. | 0 | 0 | 8 | 5 | 0
Period: Phase II - Control Extension
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation - Phase II | Control Extension - Phase II
Started | 0 | 0 | 0 | 0 | 66
Completed | 0 | 0 | 0 | 0 | 54
Not Completed | 0 | 0 | 0 | 0 | 12
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 6
Not completed — Dropped for missing two consecutive weekly safety check-ins. | 0 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Psychoeducation/Control Extension - Phase II: 5 weeks of psychoeducation about depression. Upon completion, participants will be automatically enrolled into the Limbix Spark CBT-based intervention
  Psychoeducation: The Psychoeducation program is divided into 5 lessons. Each lesson covers a different topic about depression.
  Participants who were initially assigned to the Psychoeducation control arm were given the opportunity to then complete the 5 week CBT-based intervention, Limbix Spark.
  Limbix Spark: The Limbix Spark program is divided into 5 levels. Each level provides educational information about cognitive behavioral therapy and interactive activities.
- Total: Total of all reporting groups
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation/Control Extension - Phase II | Total
Number analyzed (Participants) | 35 | 25 | 63 | 58 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 17 | 33 | 35 | 103
  Between 18 and 65 years | 17 | 8 | 30 | 23 | 78
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18 (2.36) | 17 (2.57) | 17.06 (2.49) | 16.46 (2.43) | 16.78 (2.47)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Participant Reported Gender: Female | 28 | 19 | 42 | 39 | 128
  Participant Reported Gender: Male | 6 | 5 | 16 | 10 | 37
  Participant Reported Gender: Non-Binary | 1 | 1 | 5 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 11 | 8 | 29
  Not Hispanic or Latino | 29 | 21 | 46 | 47 | 143
  Unknown or Not Reported | 0 | 0 | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2 | 4
  Asian | 7 | 4 | 4 | 0 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 2 | 10
  White | 20 | 17 | 47 | 45 | 129
  More than one race | 3 | 1 | 8 | 8 | 20
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 25 | 63 | 58 | 121

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Feasibility (Eligibility)
Description: Descriptive report of participant eligibility. Percentage of people who enrolled in each arm after expressing interest in participating in the study. Phase I participant arms are reported for this outcome.
Time Frame: Pre-enrollment
Population: People who expressed interest in participating in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Potentially Eligible Participants: The number of participants who expressed interest in participating in the study
Arm/Group | Number of Potentially Eligible Participants
Number analyzed (Participants) | 150
Participants
  Limbix Spark - Phase I | 35
  Psychoeducation - Phase I | 25

2. Primary Outcome: Number of Participants With Willingness to Participate and Program Adherence
Description: Descriptive report of willingness to participate and program adherence. Phase I participant arms are reported for this outcome.
Time Frame: From Baseline to Post Treatment (Week 5)
Population: Phase I participant arms are reported for this outcome because this was an a priori primary outcome for Phase I. Due to programming of the app, module completion was not tracked in the psychoeducation arm of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I
Number analyzed (Participants) | 35 | 25
Participants
  % of eligible participants willing to participate | 35 | 25
  % of enrolled participants completing all sessions by post-treatment: number analyzed (Participants) | 35 | 0
  % of enrolled participants completing all sessions by post-treatment | 8 |

3. Primary Outcome: Phase I - Feasibility (Satisfaction)
Description: Descriptive report of participant satisfaction (mood improvement and enjoyment) on a scale of 0-10, with 0 meaning lower satisfaction and 10 meaning higher satisfaction. Phase I participant arms are reported for this outcome.
Time Frame: Post-Treatment -"Week 5"
Population: Participants who completed the post-treatment questionnaires.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I
Number analyzed (Participants) | 24 | 18
units on a scale
  Participant Reported Mood Improvement | 5.08 (2.54) | 1.78 (2.21)
  Participant Reported Enjoyment | 6.79 (2.11) | 3.94 (2.51)

4. Primary Outcome: Phase I - Feasibility (Safety)
Description: Descriptive report of participant safety. Phase I participant arms are reported for this outcome.
Time Frame: From Baseline to Post Treatment (Week 5)
Measure: Count of Participants; unit: Participants
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I
Number analyzed (Participants) | 35 | 25
Participants
  Adverse Events | 0 | 0
  Serious Adverse Events | 0 | 2
  Adverse Device Effects | 0 | 0
  Unanticipated Adverse Device Effects | 0 | 0
  None | 35 | 23

5. Primary Outcome: Phase II - Change in Depressive Symptoms
Description: Between-subjects treatment-related change in depressive symptoms from baseline to 5-weeks as measured by Personal Health Questionnaire (PHQ-8) (min: 0; max: 24, with higher score indicating more severe depression) for those with baseline PHQ-8 ≥10.
Time Frame: Change from Baseline to Post treatment (5 weeks)
Population: Participants who had a PHQ-8 score of ≥10 at Baseline. This was a Phase II Primary Outcome measure, so only Phase II arms are reported.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Limbix Spark - Phase II | Psychoeducation - Phase II
Number analyzed (Participants) | 63 | 58
score on a scale | -5.08 [-6.72 to -3.42] | -3.51 [-5.09 to -1.93]
Statistical Analysis 1: Comparison: Limbix Spark - Phase II vs Psychoeducation - Phase II; A linear mixed-effects model (LMM) analysis was implemented on an averaged imputed dataset to evaluate main effects of Group (Spark, Control) and Week (0-5), and the Group x Week interaction. Group and Week were entered as fixed factors. Spark version, and assessment completion days since baseline were included as fixed factors to control for effects of app version and differences in time between completion of successive weekly assessments; Test type: Superiority; p = 0.06, Mixed Models Analysis; t = -1.911
Statistical Analysis 2: Comparison: Limbix Spark - Phase II vs Psychoeducation - Phase II; We used a Per Protocol approach that included participants who completed the PHQ at baseline and each week. A linear mixed-effects model (LMM) analysis was implemented on an averaged imputed dataset to evaluate main effects of Group (Spark, Control) and Week (0-5), and the Group x Week interaction; Test type: Superiority; p = 0.01, Mixed Models Analysis; t = -2.546

6. Secondary Outcome: Phase I - Change in Depression Symptoms
Description: Between-subjects treatment-related change in depressive symptoms from baseline to 5-weeks as measured by Personal Health Questionnaire (PHQ-8) (min: 0; max: 24, with higher score indicating more severe depression) for those with baseline PHQ-8 ≥5. Only Phase I participants were included in this Outcome measure.
Time Frame: From Baseline to Post Treatment (Week 5)
Population: Only Phase I participants were included in this Outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I
Number analyzed (Participants) | 34 | 23
score on a scale | -3.89 (5.29) | -3.34 (5.14)

7. Secondary Outcome: Number of Participants in Remission
Description: Remission rates based on PHQ-8 < 10 (sub-analysis for those with baseline PHQ-8 ≥ 10). Phase I and Phase II participant arms are reported for this outcome.
Time Frame: From Baseline to Post Treatment (Week 5)
Population: Participants with baseline PHQ-8 ≥ 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation/Control Extension - Phase II
Number analyzed (Participants) | 27 | 21 | 63 | 58
Participants | 13 | 7 | 11 | 2

8. Secondary Outcome: Change in Participant-rated Anxiety Symptoms and Global Functioning
Description: Between-subjects treatment-related change in participant-rated anxiety symptoms and global functioning as measured by GAD-7 Anxiety and PROMIS Pediatric Global Health Scale.
  The GAD-7 Anxiety is a brief 7-item assessment for generalized anxiety disorder. Values range from 0-21, with higher scores representing more severe anxiety.
  The PROMIS Pediatric Global Health Scale is a 7-item assessment for perceived physical, mental, and social health. Values range from 7-35, with higher scores representing better health.
  Phase I and Phase II participant arms are reported for this Outcome. Statistical Analyses are presented for Phase II results only because Phase I was intentionally not powered for analysis.
Time Frame: From Baseline to Post Treatment (Week 5)
Population: Participants who completed post-program questionnaires. Phase II participants were included if they had a baseline PHQ-8 score ≥ 10.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation/Control Extension - Phase II
Number analyzed (Participants) | 30 | 21 | 43 | 49
score on a scale
  GAD-7 | -2.87 (4.67) | -2.29 (3.94) | -3.21 (4.54) | -1.45 (3.33)
  PROMIS - General Health | 1.13 (3.64) | -0.14 (2.69) | 1.35 (3.41) | -0.35 (1.85)
Statistical Analysis 1: Comparison: Limbix Spark - Phase II vs Psychoeducation/Control Extension - Phase II; We conducted a repeated measures ANOVA (Group x Time) on GAD-7 scores to compare the change in anxiety symptoms from Baseline to Post treatment for Phase II participants who had a baseline PHQ-8 score >= 10. The interaction term is presented; Test type: Superiority; p = 0.23, ANOVA; F = 1.46
Statistical Analysis 2: Comparison: Limbix Spark - Phase II vs Psychoeducation/Control Extension - Phase II; We conducted a repeated measures ANOVA (Group x Time) on the PROMIS - General Health Score to compare the change in general health from Baseline to Post treatment for Phase II participants who had a baseline PHQ-8 score >= 10. The interaction term is reported; Test type: Superiority; p = 0.11, ANOVA; F = 2.59

9. Secondary Outcome: Change in Parent-reported Depressive Symptoms and Global Functioning.
Description: Between-subjects treatment-related change in parent-reported depressive symptoms and global functioning as measured by Mood and Feelings Questionnaire (MFQ-PS), and PROMIS Parent Proxy Global Health Scale.
  The MFQ-PS consists of a series of 13 descriptive phrases regarding how the subject has been feeling or acting in the past two weeks and is a screening tool for depression in children and young people. Values range from 0-26, with higher scores representing more severe symptoms.
  The PROMIS Parent Proxy Global Health Scale is a 7-item assessment for perceived physical, mental, and social health. Values range from 7-35, with higher scores representing better health.
  Phase I and Phase II participant arms are reported for this Outcome. Statistical Analyses are presented for Phase II results only because Phase I was intentionally not powered for analysis.
Time Frame: From Baseline to Post Treatment (Week 5)
Population: Parent/Legal Guardians of participants <18 years old who completed both baseline and post-treatment questionnaires. Phase II participants were included if they had a baseline PHQ-8 score ≥ 10.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation/Control Extension - Phase II
Number analyzed (Participants) | 10 | 8 | 23 | 27
score on a scale
  MFQ-SF | -4.20 (5.49) | -4.88 (3.60) | -4.83 (4.31) | -2.85 (4.14)
  PROMIS Parent Proxy - General Health | 0.70 (2.54) | 0.88 (2.59) | 1.21 (3.23) | 1.04 (2.47)
Statistical Analysis 1: Comparison: Limbix Spark - Phase II vs Psychoeducation/Control Extension - Phase II; We conducted a repeated measures ANOVA (Time x Group) on the MFQ to compare the change in parent report of depressive symptoms from Baseline to Post treatment for Phase II participants who had a baseline PHQ-8 score >= 10. The interaction term is presented; Test type: Superiority; p = 0.33, ANOVA; F = 0.94
Statistical Analysis 2: Comparison: Limbix Spark - Phase II vs Psychoeducation/Control Extension - Phase II; We conducted a repeated measures ANOVA (Group x Time) on the PROMIS Parent Proxy - General Health Score to compare the change in parent reported general health from Baseline to Post treatment for Phase II participants who had a baseline PHQ-8 score >= 10. The interaction term is reported; Test type: Superiority; p = 0.90, ANOVA; F = 0.02

10. Secondary Outcome: Average Treatment-related Usability and Engagement Ratings
Description: Average treatment-related usability (System Usability Scale; SUS) and engagement (User Engagement Scale-Short Form; UES-SF) ratings. Phase I and Phase II participant arms are reported for this outcome.
  The SUS is a 10-item questionnaire measuring the usability of systems. Responses range from Strongly Agree to Strongly Disagree. Scores are percentile rankings and range from 0-100. Higher scores represent higher usability.
  The UES-SF is a 12-item questionnaire measuring self-reported user-engagement. The form uses a 5-point Likert scale. Overall engagement scores range from 1-5. Higher scores represent more engagement.
Time Frame: Post-Treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation/Control Extension - Phase II
Number analyzed (Participants) | 30 | 21 | 43 | 49
units on a scale
  SUS | 80.67 (2.17) | 75.83 (2.29) | 82.85 (1.89) | 76.12 (1.92)
  UES-SF | 3.62 (0.10) | 3.10 (0.12) | 3.80 (0.08) | 3.22 (0.09)

11. Secondary Outcome: Phase II - Safety
Description: Between-group treatment-related differences in clinical concern rates and serious clinical concerns. Phase II participant arms are reported for this outcome.
Time Frame: From Baseline to Post Treatment (Week 5)
Measure: Count of Participants; unit: Participants
Arm/Group | Limbix Spark - Phase II | Psychoeducation - Phase II
Number analyzed (Participants) | 80 | 80
Participants
  Adverse Events | 4 | 2
  Serious Adverse Events | 0 | 0
  Adverse Device Effects | 0 | 0
  Unanticipated Adverse Device Effects | 0 | 0
  None | 76 | 78

12. Secondary Outcome: App Engagement and Adherence
Description: Between-group treatment-related differences in program adherence and engagement based on behavioral and mobile app analytics. Phase I and Phase II Spark participant arms are reported for this outcome. We are reporting the average number of app modules completed (out of 5 total modules).
Time Frame: From Baseline to Post Treatment (Week 5)
Measure: Mean (Standard Deviation); unit: app modules completed
Arm/Group | Limbix Spark - Phase I | Limbix Spark - Phase II
Number analyzed (Participants) | 35 | 63
app modules completed | 2.74 (1.69) | 3.17 (1.82)

ADVERSE EVENTS:
Time Frame: Adverse events were collected per patient during their 7-week (5 weeks of treatment program plus a 2 week post program questionnaire) duration of study participation. The entire duration of the study was from 30NOV2020 thru 03SEP2021.
Description: Adverse events were monitored on a daily basis via the review of free form text that could be entered by participants throughout the study and from specific questions in the weekly symptom check and weekly PHQ-8 assessments.
Arm/Group | Limbix Spark - Phase I | Psychoeducation - Phase I | Limbix Spark - Phase II | Psychoeducation - Phase II
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/25 | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/35 | 2/25 | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/35 | 0/25 | 4/80 | 2/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Limbix Spark - Phase I (N=35) | Psychoeducation - Phase I (N=25) | Limbix Spark - Phase II (N=80) | Psychoeducation - Phase II (N=80)
Hospitalized for a suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Parent reported participant hospitalization because of suicide attempt
Hospitalized for "low mood" (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Parent reported participant hospitalization for "low mood"
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Limbix Spark - Phase I (N=35) | Psychoeducation - Phase I (N=25) | Limbix Spark - Phase II (N=80) | Psychoeducation - Phase II (N=80)
Clinical Deterioration (Psychiatric disorders) | 0 | 0 | 1 | 2 — Clinical deterioration in PHQ for 2 consecutive weeks
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 2 | 0 — Participant reported suicidal ideation
Non-Suicidal Self-Injury Ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 — Parent reported that participant was experiencing Non-Suicidal Self-Injury ideation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04524598/Prot_SAP_000.pdf